CLINICAL TRIAL: NCT07095491
Title: Multidimensional Effectiveness of Self-care and Self-efficacy Based Hybrid Education in Hemodialysis Patients: A Randomised Controlled Trial on Clinical, Psychosocial and Comfort Aspects
Brief Title: Clinical, Psychosocial, and Comfort Effects of Hybrid Education in Hemodialysis Patients: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cavusoglu, Doctorate, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Mersin_University
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Interventional
Keywords: Hemodialysis; Hybrid Education; Randomized Controlled Trial; Nursing

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since hemodialysis patients participating in the study will be in either the training (experimental) or control groups, blinding will not be possible. Researchers will be blinded only during group assignment (groups A and B). Data will be transferred to a computer by the researchers, and a biostatistician independent of the study will analyze the data and report the findings, without knowing which groups A and B are assigned. This will ensure the biostatistician is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Intervention: Education group (Experimental): A structured hybrid training program based on self-care and self-efficacy will be implemented for the intervention group.
  Interventions: Other: Experimental
- Other: Control group (Other): The control group will not receive any different intervention and will continue the process with routine nursing care (standard treatment).
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — A structured hybrid training program based on self-care and self-efficacy will be implemented for the intervention group. The training will be conducted in two sessions, one day per week, over a total of two weeks.
  Arms: Experimental group: Intervention: Education group
Other: Control — The control group will not receive any different intervention and will continue the process with routine nursing care (standard treatment).
  Arms: Other: Control group

SUMMARY:
The purpose of this study is to evaluate the impact of a self-care and self-efficacy-based hybrid education program implemented for individuals receiving hemodialysis treatment on their clinical findings, psychosocial status (dialysis distress), and comfort levels during the dialysis process.

For this purpose, the most important questions to be answered in the study are as follows:

* What are the clinical findings, psychosocial status (dialysis distress), and comfort levels of hemodialysis patients at the beginning of the study?
* Does the self-care and self-efficacy-based hybrid education have an impact on the clinical findings, psychosocial status (dialysis distress), and comfort levels of hemodialysis patients?

Participants:

The intervention group will receive a structured hybrid education program based on self-care and self-efficacy. The control group will not receive any intervention during this period and will continue with routine nursing care (standard treatment).

DETAILED DESCRIPTION:
The 78 hemodialysis patients included in the study will initially be administered a personal information form, a self-care/self-efficacy scale, a hemodialysis distress thermometer, and a hemodialysis comfort scale. The intervention group will then receive a structured hybrid training program focused on self-care and self-efficacy. The training will be conducted in two sessions, one day per week, over a total of two weeks.

The training process is designed as a hybrid, incorporating both in-person and online sessions. The training will be supported by interactive sessions, practical demonstrations, guidance materials, and reminder/motivational messages sent via WhatsApp to improve individuals' self-care behaviors, psychological resilience, comfort levels, and clinical parameters.

The control group will not receive any intervention during this period and will continue with routine nursing care (standard treatment). Both groups will be assessed twice, before the training and four weeks after the training, using the relevant data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Patients who have been receiving hemodialysis treatment for at least 6 months
* Those with stable clinical findings
* Those who have not previously received professional training in self-care and self-sufficiency
* Those who have the cognitive ability to complete the data collection form
* Those who do not have a severe visual or auditory impairment
* Those who can use a smartphone and have access to the WhatsApp application
* Those who volunteer to participate in the study and sign the Informed Consent Form will be included.

Exclusion Criteria:

* Under 18 years of age
* Patients receiving hemodialysis treatment for less than 6 months
* Those whose clinical findings fluctuate to the point of being life-threatening
* Those who have previously received professional training on self-care and self-sufficiency
* Individuals who declare that they will not be able to attend at least one of the training sessions during the program
* Individuals who are simultaneously participating in another training program or psychosocial intervention
* Those who do not have the cognitive capacity to complete the data collection form
* Individuals who cannot effectively participate in the applications due to visual or hearing impairments
* Individuals who cannot use a smartphone or do not have access to the WhatsApp application
* Those who do not wish to participate in the study and who do not sign the Informed Consent Form will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Self-Care Self-Efficacy Scale | Change from before implementation and 4th week of practice
  Each item is rated on a 5-point Likert-type scale, ranging from 1 (not at all confident) to 5 (completely confident). The total score, consisting of four subscales and 10 items, ranges from 10 to 50. Higher scores indicate higher self-care and self-efficacy levels during treatment.
Haemodialysis Distress Thermometer Scale | Change from before implementation and 4th week of practice
  The scale includes a thermometer image, rated from 0 to 10. The participant indicates the overall level of distress they have felt over the past week on this scale. 0 = No distress at all, 10 = Unbearable distress. In the Turkish validation study, scores of 5 and above are generally considered clinical distress.
Hemodialysis Comfort Scale | Change from before implementation and 4th week of practice
  The scale, consisting of two subscales, is rated on a 5-point Likert-type scale (1 = never, 5 = always). The total score from the scale ranges from 9 to 45. Higher scores indicate a higher level of comfort for the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çavuşoğlu, Doctorate, Study Director — Mersin University; Esra Köse, Doctorate, Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No